CLINICAL TRIAL: NCT03256461
Title: Multi-center Clinical Trial of Lactate Clearance Goal-directed Fluid Resuscitation in Patients With Sepsis
Brief Title: Lactate Clearance Goal-directed Therapy in Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LCGRIS-01
Record Dates: First submitted 2017-08-07; First posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Sepsis
Keywords: sepsis; lactate clearance; protocolized resuscitation
MeSH Terms: conditions — Sepsis | interventions — Lactase; Population Groups

STUDY DESIGN:
Intervention Model Description: This trial is a prospective, multicenter, single-blind, parallel-group, central-randomized, controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lactate clearance 10% target group (Experimental): Lactate clearance falls by 10-percent every two hours.
  Interventions: Behavioral: Lactate clearance 10% target group
- Lactate clearance 20% target group (Experimental): Lactate clearance falls by 20-percent every two hours.
  Interventions: Behavioral: Lactate clearance 20% target group
- Standard EGDT group (Placebo Comparator): Refer to the Surviving Sepsis Campaign(SSC) 2012 sepsis guidelines within 6 h liquid resuscitation.
  Interventions: Behavioral: Standard EGDT group

INTERVENTIONS:
Behavioral: Lactate clearance 10% target group — Participants receive the protocolized resuscitation to achieve the goal of 10-percent lactate clearance every two hours within the initial six hours of treatment.
  Other Names: Lac% 10% group
  Arms: Lactate clearance 10% target group
Behavioral: Lactate clearance 20% target group — Participants receive the protocolized resuscitation to achieve the goal of 20-percent lactate clearance every two hours within the initial six hours of treatment.
  Other Names: Lac% 20% group
  Arms: Lactate clearance 20% target group
Behavioral: Standard EGDT group — Participants receive the strategy of early goal-directed treatment of sepsis fluid resuscitation.
  Other Names: EGDT group
  Arms: Standard EGDT group

SUMMARY:
Serum lactate level is depended on the balance between lactate production and clearance. It is seen as a sensitive indicator reflecting not only the low systemic perfusion but microcirculatory dysfunction which cause global or regional tissue hypoxia (as a result of impaired mitochondrial oxidation). 2016 Surviving Sepsis Campaign guideline stated "We suggest guiding resuscitation to normalize lactate in patients with elevated lactate levels as a marker of tissue hypoperfusion", with weak recommendation and low quality of evidence. Several trials which evaluated the resuscitation strategy included lactate clearance as a target while based on 2.0 diagnostic criteria for sepsis, finally showed conflicting results. The aim of this study is to explore the feasibility of lactate clearance guide resuscitation in sepsis that defined by The Third International Consensus Definitions for Sepsis and Septic shock through multi-center, central-randomization clinical trial.

DETAILED DESCRIPTION:
Sepsis remains a great challenge for clinicians, early goal-directed therapy(EGDT), referring to a number of target-achieving indicators including systemic central venous oxygen saturation(ScvO2) after initial fluid resuscitation within 6 hours, has been one of the main treatment for sepsis. ScvO2 is the only indicator that reflects tissue oxygen metabolism. However, there're studies confirmed that ScvO2 oriented EGDT cannot reduce the mortality of sepsis. So it is important to find out a more effective indicator. Lactic acid is a product of anaerobic metabolism of the body, lactate clearance has been found to effectively predict the prognosis of sepsis. Few studies have shown that lactate clearance oriented fluid resuscitation can be of benefit in patients with sepsis. Nevertheless, whether lactate clearance could be combined with sepsis Bundle as a new marker to improve the prognosis remains a problem. The objective of this study is to discuss the feasibility of lactate clearance oriented sepsis treatment through multi-center clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Older than 17 years old.
* Primary diagnosis is sepsis, means being confirmed or suspected infection while have at least 2 points of quickSOFA(qSOFA).
* Be transferred to intensive care unit (ICU) for the first time during this hospitalization.
* Elevated lactate ≥3.0mmol/L.

Exclusion Criteria:

* Acute hemorrhage uncontrolled.
* Pregnancy.
* Known liver disease - Child-Pugh classes C, acute hepatic failure, severe hepatopathy accompany with prominent portal hypertension.
* Known being in an immunosuppressive state:

  1. Suffering from any disease that is unrelated with sepsis that severely inhibits the immune to infection, such as: active hematological or lymphoma malignancy, or during immunosuppressive therapy, such as chemotherapy or radiotherapy.
  2. Known human immunodeficiency virus (HIV) serology positive.
* Known chronic kidney disease.
* Suffering from any disease that affects lactate kinetics, such as mitochondrial encephalopathy, congenital hyperlipidemia, Wernicke encephalopathy, etc. Or other probable cause of hyperlactatemia.
* Took any drugs that affect lactate kinetics within the effective time window, such as taking metformin or phenylephrine within 1 week.
* Suffering from any disease that restricts resuscitation, such as heart failure, cardiac surgery, severe heart disease etc, or suffered from a cardio-pulmonary resuscitation,.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1128 (Estimated)
Dates: Start 2017-08-21 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
28-d mortality | Four years
  All-cause mortality at 28 days

SECONDARY OUTCOMES:
ICU Length of stay | Four years
  Length of stay in the intensive care unit (ICU)
Hospital Length of stay | Four years
  Length of stay in hospital
90-d mortality | Four years
  All-cause mortality at 90 days
In-hospital mortality | Four years
  All-cause mortality during hospitalization
In-ICU mortality | Four years
  All-cause mortality during ICU stay
Administered treatments | Four years
  Administered treatments included: crystalloid volume, vasopressor administered, dobutamine, red blood cell(RBC) transfusion, mechanical ventilation, renal-replacement therapy
SOFA at 24h | Four years
  Sequential Organ Failure Assessment(SOFA) at 24 hours
Adverse events | Four years
  Proportion of patients reporting treatment-emergent adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Chen Zhongqing, Ph.D, Study Chair — Southern Medical University
Locations (1):
- NanFang hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT03256461/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT03256461/ICF_001.pdf